CLINICAL TRIAL: NCT02576756
Title: Retrospective Study of the Risk of Aspiration and Postoperative Pulmonary Problems in Patients Who Have Had a Difficult Intubation.
Brief Title: Retrospective Study in Patients Who Have Had a Difficult Intubation.
Status: Completed | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Other Study IDs: PULINT
Record Dates: First submitted 2015-10-13; First posted 2015-10-15 (Estimated); Last update posted 2025-11-18 (Actual); Status verified 2016-08

CONDITIONS: Aspiration; Pneumonia
Keywords: Risk on aspiration; Postoperative; Difficult Intubation
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- with difficult intubation: Control population
- without difficult intubation: Control population

SUMMARY:
The investigator wants to investigate if there is an increased risk of postoperative pulmonary problems in patients who have had an intubation where there was need for more than a laryngoscope.

DETAILED DESCRIPTION:
A difficult intubation is defined as an intubation in which more than a laryngoscope was needed.

Afterwards patient data retrieved from the Clinical Work Station: age, type of operation and time, date, type of anaesthesia, de tools needed for intubation, time needed for intubation and anaesthesia.

In the Clinical Work Station of the Hospital the investigator will search for the following data in these selected patients: preoperative comorbidities, home medication, type of postoperative pulmonary problems and the treatment that was given, time of hospital stay and which department the patient stayed.

Patients with a difficult intubation will be linked to a patient with a corresponding medical history and type of operation but without a difficult intubation. The investigator will look for the same parameters of these patients in the Clinical Work Station.

By means of an odds-ratio the relative risk of a pulmonary complication after a difficult intubation in connection with an easy intubation with different variables can be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Every patient who had an intubation where another device than a laryngoscope was necessary

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Every patients who had an intubation where another device than a laryngoscope was necessary
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Relative risk for postoperative pulmonary incidents | 6 months
  number of participants with Relative risk

CONTACTS AND LOCATIONS:
Overall Officials: Josia B Glissenaar, Med student, Principal Investigator — Universitair Ziekenhuis Brussel; Jan Poelaert, PhD MED, Study Chair — Universitair Ziekenhuis Brussel

IPD SHARING:
Plan to Share IPD: No